CLINICAL TRIAL: NCT00110058
Title: A Multi-Center Phase II Study of Nonmyeloablative Conditioning With TBI and Fludarabine for HLA-Matched Related Hematopoietic Cell Transplantation for Treatment of Chronic Myeloid Leukemia in Chronic and Accelerated Phase
Brief Title: Fludarabine and Radiation Therapy in Treating Patients Who Are Undergoing Donor Stem Cell Transplant for Chronic Phase or Accelerated Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1954.00; FHCRC-1954.00; CDR0000423314 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interferon-alpha; Cyclosporine; fludarabine phosphate; Imatinib Mesylate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: imatinib mesylate
Drug: mycophenolate mofetil
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and radiation therapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) or interferon alfa after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine together with radiation therapy works in treating patients who are undergoing donor stem cell transplant for chronic phase or accelerated phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the disease-free survival rate in patients with chronic or accelerated phase chronic myelogenous leukemia that failed or inadequately responded to prior imatinib mesylate treated with nonmyeloablative conditioning comprising fludarabine and low-dose total-body irradiation followed by allogeneic peripheral blood stem cell transplantation.

Secondary

* Determine the complete cytogenetic and molecular response rates in patients treated with this regimen.
* Determine overall survival of patients treated with this regimen.
* Determine non-relapse mortality in patients treated with this regimen.
* Determine the incidence of serious infection, graft-versus-host disease, and myelosuppression in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Conditioning treatment: Patients receive fludarabine IV on days -4 to -2. Patients undergo low-dose total-body irradiation (TBI) on day 0.
* Allogeneic peripheral blood stem cell transplantation: After TBI, patients undergo allogeneic peripheral blood stem cell transplantation on day 0.
* Immunosuppression: Patients receive oral cyclosporine twice daily on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease (GVHD). Patients also receive oral mycophenolate mofetil twice daily on days 0-27.
* Post-transplant treatment: Patients experiencing disease persistence or progression AND low donor chimerism discontinue immunosuppression. Patients with disease persistence or progression after discontinuing immunosuppression receive oral imatinib mesylate once daily. Patients who have disease improvement after day 28 of imatinib mesylate treatment AND who have no evidence of disease after day 84 of imatinib mesylate treatment continue imatinib mesylate in the absence of disease progression or unacceptable toxicity. Patients who fail to improve after day 28 of imatinib mesylate treatment OR who have residual disease after day 84 of imatinib mesylate treatment receive donor lymphocytes IV over 15-30 minutes once every 1-4 months for up to 4 infusions. Patients ineligible to receive donor lymphocytes (e.g., patients with evidence of GVHD) receive interferon alfa subcutaneously 3 times a week for up to 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 6, 9, 12, 18, and 24 months, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Philadelphia chromosome-positive (Ph+) chronic myelogenous leukemia, meeting 1 of the following criteria:

  * Chronic phase

    * Ph+ by cytogenetics or fluorescent in situ hybridization (FISH) assay
  * Accelerated phase, meeting any of the following criteria:

    * More than 10% but < 30% myeloblasts and promyelocytes in marrow or peripheral blood
    * Any additional clonal cytogenetic abnormalities
    * Increasing splenomegaly
    * Extramedullary tumor
    * WBC, platelet count, or hematocrit perturbations not controlled by therapy with hydroxyurea, interferon, or imatinib mesylate
    * Persistent unexplained fever or bone pain
* Less than 5% blasts in the marrow at time of transplantation
* Not eligible for OR refused conventional myeloablative allogeneic stem cell transplantation
* Failed OR suboptimal response to prior imatinib mesylate, as defined by 1 of the following:

  * Absence of complete hematologic response after > 3 months of treatment with imatinib mesylate
  * Absence of cytogenetic response, as defined by 1 of the following:

    * Absence of any cytogenetic response (< 95% Ph+ or BCR/ABL+ cells by cytogenetic or FISH analysis, respectively) after 6 months of treatment with imatinib mesylate
    * Absence of major cytogenetic response (< 35% Ph+ or BCR/ABL+ cells by cytogenetic or FISH analysis, respectively) after 1 year of treatment with imatinib mesylate
    * Absence of complete cytogenetic response (no Ph+ cells by cytogenetic analysis OR BCR/ABL+ cells within normal limits by FISH analysis) after 18 months of treatment with imatinib mesylate
  * Hematologic evidence of disease progression
  * Cytogenetic evidence of disease progression

    * Increase in Ph+ cells or BCR/ABL+ cells by > 20% with at least 1 month between sequential testing
  * Molecular evidence of disease progression

    * More than 10-fold increase in BCR/ABL mRNA levels by quantitative polymerase chain reaction (Q-PCR) with at least 1 month between 2 sequential tests
  * Experienced adverse events during treatment with imatinib mesylate that precluded further administration of the drug
* No CNS disease refractory to intrathecal chemotherapy
* HLA identical related donor available

  * Phenotypically matched at HLA-A, -B, -C, DRQ1, and DBQ1
* No presence of circulating leukemic blasts by standard pathology

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Karnofsky 70-100% OR
* Lansky 70-100%

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* No fulminant liver failure
* No cirrhosis of the liver with evidence of portal hypertension or bridging fibrosis
* No alcoholic hepatitis
* No esophageal varices
* No history of bleeding esophageal varices
* No hepatic encephalopathy
* No uncorrectable hepatic synthetic dysfunction evidenced by prolongation of PT
* No ascites related to portal hypertension
* No bacterial or fungal liver abscess
* No biliary obstruction
* No chronic viral hepatitis AND bilirubin > 3 mg/dL
* No symptomatic biliary disease

Renal

* Renal failure allowed

Cardiovascular

* No symptomatic coronary artery disease
* Ejection fraction ≥ 35%
* No other cardiac failure requiring therapy
* No poorly controlled hypertension (blood pressure ≥ 150/90 mm Hg) on standard medication

Pulmonary

* DLCO ≥ 30%
* Total lung capacity ≥ 30%
* FEV_1 ≥ 30%
* No requirement for continuous supplementary oxygen
* No fungal pneumonia with radiological progression after treatment with amphotericin or mold-active azoles for > 1 month

Other

* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for 12 months after completion of study treatment
* HIV negative
* No other disease that severely limits life expectancy
* No other active malignancy except localized nonmelanoma skin cancer
* No nonhematologic malignancy within the past 5 years that is currently in complete remission and has a > 20% risk of disease recurrence except for nonmelanoma skin cancer
* No systemic uncontrolled infection
* No active bacterial or fungal infection unresponsive to medical therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 48 hours since prior imatinib mesylate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-02; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Rate of complete molecular response
Late nonrelapse mortality
Incidence and severity of graft-vs-host disease (GVHD)
Incidence of serious infections
Myelosuppression
Overall survival and disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241